CLINICAL TRIAL: NCT03116360
Title: Comparison of Ultrasound and X-ray as Screening Tests for Diagnosis of Lower Extremity Stress Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Virginia (Other)
Collaborators: NBA&GE Orthopedics and Sports Medicine Collaboration (Unknown)
Responsible Party: Principal Investigator, David Hryvniak, MD, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 19779
Record Dates: First submitted 2017-04-07; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Stress Fracture; Ultrasound Therapy; Musculoskeletal Ultrasound
MeSH Terms: conditions — Fractures, Stress | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Subjects suspected to have an acute stress fracture of the lower extremity will be recruited. Subjects will be required to have already undergone the initial step of the traditional diagnostic algorithm with x-ray as part of clinical care of the suspicious region on the day of enrollment. A physical exam and vital signs will be obtained as part of standard clinical care. All subjects will then be scheduled to undergo diagnostic ultrasound for research purposes at a separate appointment with ultrasound procedure performed by a blinded clinical physician boarded in Physical Medicine and Rehabilitation, competent in performing and reading diagnostic ultrasound. All subjects will then undergo a confirmatory MRI without contrast of the region of concern. The MRI may be ordered as part of clinical care or for research if not required for clinical purposes. MRI screening per standard processes will be done by the MRI staff.
Masking Description: Subjects will be required to have already undergone the initial step of the traditional diagnostic algorithm with x-ray of the suspicious region. All subjects will then be scheduled to undergo diagnostic ultrasound at a separate appointment with ultrasound procedure performed by a blinded clinical physician. All patients will then undergo a confirmatory MRI of the region of concern. A statistician in the Department of Public Health at the University of Virginia will be performing statistical analysis. All x-ray and MRI obtained for this study will be read by a Radiologist board certified in Musculoskeletal Radiology. Diagnostic ultrasound performance: The physician performing the ultrasound will be blinded to the results of the x-ray and MRI. The physician performing the ultrasound will be informed of the bone in question (ex. Tibia) and will be able to perform a focused history and exam.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): All patients will undergo traditional xray screening as well as experimental screening with diagnostic ultrasound. All subjects will undergo confirmatory MRI.
  Interventions: Diagnostic Test: Diagnostic Ultrasound

INTERVENTIONS:
Diagnostic Test: Diagnostic Ultrasound — The physician performing the ultrasound will be blinded to the results of the x-ray and MRI. The physician performing the ultrasound will be informed of the bone in question (ex. Tibia) and will be able to perform a focused history and exam. The bone in which acute stress fracture is suspected will then be scanned throughout its length in two orthogonal views. The criteria for diagnosing acute stress fracture on ultrasound include displaying 2 out of 3 of the following: hypoechoic periosteal elevation of cortical bone, visible cortical disruption, hyperemia surrounding the periosteal lesion on power Doppler. The ultrasound physician will then be asked to make a determination whether the ultrasound study is positive for acute stress fracture or negative/indeterminate.

SUMMARY:
Hypothesis: Diagnostic ultrasound is an appropriate screening test for acute stress fracture in the lower extremity and is superior to x-ray.

Primary Aims: To determine if diagnostic ultrasound is an appropriate screening test with high sensitivity and at least moderate specificity for the identification of acute stress fractures of the lower extremity.

Methods: In this double-blind, prospective clinical study, subjects (age 14 years and up) suspected to have an acute stress fracture of the lower extremity will be recruited from the Sports Medicine clinic at the University of Virginia Health System in the Department of Physical Medicine & Rehabilitation. Subjects will undergo the traditional diagnostic algorithm including screening x-ray as part of standard care. Subjects will then undergo a confirmatory MRI of the region of concern if the initial x-ray was negative as part of standard care. Any subject who does not require an MRI for clinical purposes (initial X-ray was positive) will have one completed for research purposes. All subjects will also undergo diagnostic ultrasound performed by a separate, blinded physician competent in diagnostic ultrasound for research purposes. A statistician in the Department of Public Health at the University of Virginia will be performing statistical analysis during data analysis. Findings will be analyzed using a McNemar chi-square test to evaluate for significant differences between the sensitivities of ultrasound and x-ray.

DETAILED DESCRIPTION:
Primary aims: To determine if diagnostic ultrasound is an appropriate screening test (high sensitivity and at least moderate specificity) and non-inferior to x-ray for diagnosis of acute stress fracture of the lower extremity.

Secondary Aims: To determine what grade(s) of acute stress fracture that x-ray and ultrasound are capable of detecting reliably and accurately.

Population: Subjects will be recruited from the Sports Medicine clinic at the University of Virginia Health System in the Department of Physical Medicine and Rehabilitation. Subjects will have suspected acute stress fracture of the lower extremity and will be age 14 years and older. Anatomic locations included in this study are as follows: all bones of the foot and ankle, tibia, fibula, and femoral shaft. Patients with suspected stress fracture of the femoral neck will be excluded due to the difficulty of appropriate ultrasound evaluation secondary to depth as well as the potential for significant morbidity if not diagnosed properly. We estimate that the Sports Medicine clinic diagnoses approximately 12 acute stress fractures per month per physician amongst the three physician's clinics involved in this study. Therefore, our anticipated number of subjects over a 6 month period will be at least 216 patients.

Design: In this double-blind , prospective clinical study, subjects suspected to have an acute stress fracture of the lower extremity will be recruited from Sports Medicine Clinic (conducted by two physicians boarded in Physical Medicine and Rehabilitation and one physician board in Family Medicine and all boarded in Sports Medicine). When patients present to one of three physicians in Sports Medicine Clinic with a suspected acute stress fracture of the lower extremity, they will be offered the opportunity to enroll. Subjects will be required to have already undergone the initial step of the traditional diagnostic algorithm with x-ray of the suspicious region on the day of enrollment. All subjects will then be scheduled to undergo diagnostic ultrasound at a separate appointment with ultrasound procedure performed by a blinded clinical physician boarded in Physical Medicine and Rehabilitation, competent in performing and reading diagnostic ultrasound. All patients will then undergo a confirmatory MRI of the region of concern. Subject recruitment and data collection are expected to be completed over a six-month period. A statistician in the Department of Public Health at the University of Virginia will be performing statistical analysis. We plan to analyze findings using a McNemar chi-square test to evaluate for significant differences between the sensitivities of ultrasound and x-ray in diagnosing acute stress fracture of the lower extremity. All x-ray and MRI obtained for this study will be read by a Radiologist board certified in Musculoskeletal Radiology.

Diagnostic ultrasound performance: The physician performing the ultrasound will be blinded to the results of the x-ray and MRI. The physician performing the ultrasound will be informed of the bone in question (ex. Tibia) and will be able to perform a focused history and exam. The bone in which acute stress fracture is suspected will then be scanned throughout its length in two orthogonal views. The criteria for diagnosing acute stress fracture on ultrasound include displaying 2 out of 3 of the following: hypoechoic periosteal elevation of cortical bone, visible cortical disruption, hyperemia surrounding the periosteal lesion on power Doppler. The ultrasound physician will then be asked to make a determination whether the ultrasound study is positive for acute stress fracture or negative/indeterminate.

Statistical Analysis/Power Analysis: Sensitivity and specificity of diagnostic ultrasound and x-ray were calculated. MRI was used as the gold standard confirmatory test. Positive predictive value and Negative predictive value were also calculated for comparison. A priori power analysis determined a sample size of 186 was needed to obtain a power of 80%. The primary aim will be analyzed using a bootstrap test to compare the x-ray sensitivity to the ultrasound sensitivity. In order to account for the paired nature of the data, the bootstrap sampling will be at the subject level and will draw pairs with the x-ray and ultrasound outcomes associated with individual subjects. A statistician from the University of Virginia was hired for all statistical calculations.

Subject Recruitment: Subjects presenting to the Sports Medicine clinic with suspected acute stress fracture of the lower extremity on initial presentation will be offered participation. Participation includes an additional clinic visit with a separate physician to perform a diagnostic ultrasound of the area of concern in addition to the standard work up they would receive for their presenting complaint. Informed consent was obtained at the time of study enrollment. Subjective will be offered ultrasound evaluation as well as follow up confirmatory MRI. The cost of follow up MRI is included in the study to prevent selection bias based on insurance coverage for MRI. The costs associated with the additional clinic visit for diagnostic ultrasound is also included in the study budget.

ELIGIBILITY:
Inclusion Criteria:

* age 14 years and up
* suspected acute stress fracture of the lower extremity
* symptoms < 4 weeks
* x-ray ordered by clinician to which subjects originally present with suspected stress fracture

Exclusion Criteria:

* age < 14
* unable to provide consent
* unable to undergo MRI (implantable pacemaker or other device not compatible for MRI)
* previous diagnosis of acute stress fracture in the location of interest
* previous XR or MRI obtained at an outside clinic/facility prior to presentation
* previously implanted hardware (ex. orthopedic screws or plates) at location of interest
* symptoms > 8 weeks
* depth from skin surface to bone surface that exceeds the capability of ultrasound for visualization
* Pregnant (self-reported)
* Subject is known to all clinicians who would be completing the diagnostic ultrasound component of the study
* Open wound at site of suspected stress fracture

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority comparison of diagnostic ultrasound to x-ray | 6 months
  Comparison of sensitivity between diagnostic ultrasound and x-ray for acute stress fractures of the lower extremity.

SECONDARY OUTCOMES:
Comparing ultrasound and x-ray across severity of stress fracture | 6 months
  Comparison of sensitivity and accuracy of diagnostic ultrasound and x-ray stratified across MRI grading of acute stress fracture of the lower extremity.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khy V, Wyssa B, Bianchi S. Bilateral stress fracture of the tibia diagnosed by ultrasound. A case report. J Ultrasound. 2012 Jun;15(2):130-4. doi: 10.1016/j.jus.2011.09.002. Epub 2011 Sep 16. PMID 23396635
- [Background] Nitz AJ, Scoville CR. Use of ultrasound in early detection of stress fractures of the medial tibial plateau. Mil Med. 1980 Dec;145(12):844-6. No abstract available. PMID 6779231
- [Background] Uri Farkash et al. Ultrasonography as a diagnostic modality of tibial stress fractures. J Musculoskelet Res. 11, 55 (2008).
- [Background] Romani WA, Perrin DH, Dussault RG, Ball DW, Kahler DM. Identification of tibial stress fractures using therapeutic continuous ultrasound. J Orthop Sports Phys Ther. 2000 Aug;30(8):444-52. doi: 10.2519/jospt.2000.30.8.444. PMID 10949501
- [Background] Papalada A, Malliaropoulos N, Tsitas K, Kiritsi O, Padhiar N, Del Buono A, Maffulli N. Ultrasound as a primary evaluation tool of bone stress injuries in elite track and field athletes. Am J Sports Med. 2012 Apr;40(4):915-9. doi: 10.1177/0363546512437334. Epub 2012 Feb 23. PMID 22366519
- [Background] Boam WD, Miser WF, Yuill SC, Delaplain CB, Gayle EL, MacDonald DC. Comparison of ultrasound examination with bone scintiscan in the diagnosis of stress fractures. J Am Board Fam Pract. 1996 Nov-Dec;9(6):414-7. PMID 8923399
- [Background] Banal F, Gandjbakhch F, Foltz V, Goldcher A, Etchepare F, Rozenberg S, Koeger AC, Bourgeois P, Fautrel B. Sensitivity and specificity of ultrasonography in early diagnosis of metatarsal bone stress fractures: a pilot study of 37 patients. J Rheumatol. 2009 Aug;36(8):1715-9. doi: 10.3899/jrheum.080657. Epub 2009 Jun 30. PMID 19567620
- [Background] Battaglia PJ, Kaeser MA, Kettner NW. Diagnosis and serial sonography of a proximal fifth metatarsal stress fracture. J Chiropr Med. 2013 Sep;12(3):196-200. doi: 10.1016/j.jcm.2013.10.002. PMID 24396321
- [Background] Wright AA, Hegedus EJ, Lenchik L, Kuhn KJ, Santiago L, Smoliga JM. Diagnostic Accuracy of Various Imaging Modalities for Suspected Lower Extremity Stress Fractures: A Systematic Review With Evidence-Based Recommendations for Clinical Practice. Am J Sports Med. 2016 Jan;44(1):255-63. doi: 10.1177/0363546515574066. Epub 2015 Mar 24. PMID 25805712
- [Background] Starkey C. Injuries and illnesses in the national basketball association: a 10-year perspective. J Athl Train. 2000 Apr;35(2):161-7. PMID 16558626
- [Background] Taylor PM, Gordon G, Lowe MK: Basketball injuries. In: Subotnik SI (ed): Sports Medicine of the Lower Extremity (2nd edition), Ch. 31, W.B. Saunders Co., Philadelphia, 1999, p. 695.
- [Background] Bennell KL, Malcolm SA, Thomas SA, Wark JD, Brukner PD. The incidence and distribution of stress fractures in competitive track and field athletes. A twelve-month prospective study. Am J Sports Med. 1996 Mar-Apr;24(2):211-7. doi: 10.1177/036354659602400217. PMID 8775123
- [Background] Brudvig TJ, Gudger TD, Obermeyer L. Stress fractures in 295 trainees: a one-year study of incidence as related to age, sex, and race. Mil Med. 1983 Aug;148(8):666-7. No abstract available. PMID 6415522
- [Background] Strowbridge NF. Musculoskeletal injuries in female soldiers: analysis of cause and type of injury. J R Army Med Corps. 2002 Sep;148(3):256-8. doi: 10.1136/jramc-148-03-06. PMID 12469426
- [Background] Liong SY, Whitehouse RW. Lower extremity and pelvic stress fractures in athletes. Br J Radiol. 2012 Aug;85(1016):1148-56. doi: 10.1259/bjr/78510315. PMID 22815414
- [Background] Moran DS, Evans RK, Hadad E. Imaging of lower extremity stress fracture injuries. Sports Med. 2008;38(4):345-56. doi: 10.2165/00007256-200838040-00005. PMID 18348592